CLINICAL TRIAL: NCT04045574
Title: DAMP1: The 1T1T Concept Versus Conventional Implant Loading Protocol: A Comparative Study
Brief Title: DAMP1: The 1T1T Concept Versus Conventional Implant Loading Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Mainjot Amélie, Clinical Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA001
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Dental Implant Failure; Dental Prosthesis Failure
Keywords: CAD-CAM system; Immediate dental implant loading; PICN; Comparative study

STUDY DESIGN:
Intervention Model Description: single center comparative controlled trials
Masking Description: the technique to be used for each site will be randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAMP1 : (Experimental): Single arm trial comparing a conventional technique with an experimental one, within the same patient.
  Interventions: Procedure: The 1T1T concept versus conventional implant loading protocol

INTERVENTIONS:
Procedure: The 1T1T concept versus conventional implant loading protocol — Implant placement followed by either a conventional or a delayed loading of a PICN screw-retained crown.

SUMMARY:
The One tooth - One time (1T1T) innovative approach is a straightforward and cost-effective protocol to replace a missing tooth in the posterior region (Lambert and Mainjot 2017) (see Appendix). The digital impression of single unit implants right after the implant placement and the direct manufacturing of a Polymer-Infiltrated Ceramic Network (PICN) screw-retained crown allows the delivery of a final tooth in occlusion within the same day. The absence of lab procedures reduces the number of appointments, providing immediate results and high patient satisfaction. The prosthesis material choice is crucial in this procedure. Indeed, PICN high resilience, i.e. damping effect, could reduce peri-implant strain compared to ceramic materials (Magne, Silva et al. 2013) (Maminskas, Puisys et al. 2016), moreover its elastic modulus is close to tooth tissues, while other CAD-CAM composites value is too low and ceramic materials are too high. The rapid milling and manufacturing process, without any firing procedure, and the ease of adjustments (particularly to adjust proximal and occlusal contact points), make also PICNs well-adapted to chair-side systems. The material low stiffness and hardness can improve patient comfort and promote adaptation of the restorations to occlusal relationships with time. The 1T1T approach was presented as a proof of concept in a first international publication using tissue level implants from Straumann, which describes the whole protocol (Lambert and Mainjot 2017). Currently, a case series including 10 teeth is on-course, showing a 100% survival rate of implants and restorations after a 2-yr follow-up. These results are very promising but further clinical research is needed to validate such a protocol on a larger number of patients, on other implant systems as well as to compare this approach to conventional protocols.

DETAILED DESCRIPTION:
The present study is designed as a single center comparative controlled trial. This study aims to compare immediate (1T1T) versus delayed loading with a final PICN screw-retained crown (DL-PICN), performed with CAD-CAM system. A total of 28 consecutive patients (56 teeth) above the age of 18 and presenting two single-unit edentulous space in the posterior region (molars or premolars, upper or lower jaw), will be considered for possible inclusion in the study, according to the inclusion and exclusion criteria (patients with high occlusal stress will be included).

The performance of the different protocols will be tested in terms of (1) prostheses and implants survival and success rates following international standards (2) Patient reported outcome measures (PROMs); (3) time and cost. Moreover, restorations and antagonistic teeth wear will be studied trough ex-vivo analysis by profilometry of replica. The evaluations will be carried out at a follow-up period of 7 days, 2, 6 months and then every year up to 5 years.

Hypothesis is that the type of loading technique with a final PICN crown (1T1T or DL-PICN) does not influence prostheses and implants survival and success rates, but that 1T1T protocol improves patient-centered outcomes as well as time and cost effectiveness in comparison with DL-PICN.

The overall cost of the restoration treatment will be 1600€ (instead of 2100€), which represents a saving of 500€ for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have voluntarily signed the informed consent form before any study related action
* Age : 18 or above
* Men/Women
* Patient in good systemic health (ASA I/ II)
* No contraindication against oral surgical interventions
* Full mouth plaque score (FMPI) lower or equal than 25%
* Patient with two single unit edentulous space in the posterior area, upper or lower jaw, seeking for implant therapy
* Maximum two missing teeth per quadrant
* Two single unit edentulous spaces can be contiguous if there are three posterior teeth in occlusal contact in the tested half arch.
* After the crown placement, at least 3 posterior teeth must be in occlusal contact with the antagonistic teeth in the tested half arch.
* The tooth at the implant site must have been extracted or lost at least 12 weeks before the date of implantation.
* At least 8 mm of bone in the vertical dimension
* At least 6 mm of bone in the bucco-lingual dimension.

Exclusion Criteria:

* Autoimmune disease requiring medical treatment
* Medical conditions requiring prolonged use of steroids
* Use of Bisphosphonate intravenously or more then ˃ 3 years of oral use
* Infection (local or systemic) - patient with gingivitis or active local infection will undergo a medical treatment prior to his entrance to the study, each individual will be evaluated prior to study procedure for suitability, in case of systemic infection the evaluation will be based on medical anamneses, and if necessary will be referred to relevant medical tests.
* Current pregnancy or breastfeeding women
* Alcoholism or chronically drug abuse
* Immunocompromised patients
* Uncontrolled Diabetes
* Smokers (more than 10 cigarettes/day)
* Prisoners
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Prostheses survival/success rates following international standards | up to 5 years
Implants survival/success rates following international standards | up to 5 years
Patient reported outcome measures (PROMs) | up to 5 years
  Questionnaires will be used to assess outcome measure
Time of protocols | up to 2 months
Cost of protocols | up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Dentistry University of Liege, Liège, Choose A State, Belgium

IPD SHARING:
Plan to Share IPD: No